CLINICAL TRIAL: NCT07027267
Title: A Prospective, Multi-Center, Open-Label Study to Evaluate the Safety and Effectiveness of TurbAlign™ to Achieve Middle Turbinate Medialization After Functional Endoscopic Sinus Surgery (FESS) (GAIA)
Brief Title: Safety and Effectiveness of TurbAlign™ for Middle Turbinate Medialization After Functional Endoscopic Sinus Surgery
Acronym: Gaia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spirair, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-004
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Sinus Endoscopic Surgery; Turbinate
Keywords: Sinus surgery; FESS; middle turbinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Open-label (Experimental): Treatment with the Spirair device as a treatment for medialization of the middle turbinates
  Interventions: Device: Implantation of Spirair device into the middle turbinates; Device: TurbAlign

INTERVENTIONS:
Device: Implantation of Spirair device into the middle turbinates — The Spirair implant is designed to separate the middle turbinate from the lateral nasal wall during the healing phase associated with nasal/sinus surgery.
  Other Names: TurbAlign
Device: TurbAlign — The Spirair implant is designed to separate the middle turbinate from the lateral nasal wall during the healing phase associated with nasal/sinus surgery

SUMMARY:
A study of a bioabsorbable implant to separate the middle turbinate from the lateral nasal wall associated with nasal/sinus surgery

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of the Spirair implant as a primary treatment to achieve medialization of the middle turbinate after functional endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 to ≤ 70 years of age at time of consent
* Subject scheduled to undergo bilateral endoscopic sinus surgery
* Able to speak, read and understand English
* Willing and able to provide informed consent and comply with the study protocol

Exclusion Criteria:

* History of removal of one or both middle turbinates
* Presence of significant concha bullosa, which requires surgical excision
* Presence of non-viable tissue at the implantation site
* Active infection at the implantation site
* Chronic nasal decongestant use (i.e. Afrin, etc)
* Recreational intra-nasal drug use within 12 months of enrollment
* Documented evidence of a history (e.g., liver testing) of drug/alcohol abuse within 12 months of enrollment
* Hypersensitivity to any investigational device materials including known or suspected allergy to poly(dioxanone) (PDO) or other bioabsorbable materials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Miller Synechia Score | 8 Weeks
  Rate of lateral synechia formation resulting in occlusion of the middle meatus at each turbinate (Miller Synechia Score of 2 or 3) observed at 8 weeks.

SECONDARY OUTCOMES:
Middle Turbinate Position Grade | 4 and 8 weeks
  Rate of avoidance of the middle turbinate lateralization at 4 and 8 weeks using Middle Turbinate Position Grade
Miller Synechia Score | 4 weeks
  Rate of lateral synechia formation resulting gin occlusion of the middle meatus at each turbinate (Miller Synechia Score of 2 or 3) observed at 4 weeks
Inflammation assessment | 8 weeks
  Inflammation assessment of the gross tissue appearance at implantation site is assessed via live endoscopic video and graded I: None, II: Mild, III: Moderate, IV: Severe by investigator at 8 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - LSU Health Science Center, Shreveport, Louisiana
  - Houston Methodist ENT Specialists, Houston, Texas

IPD SHARING:
Plan to Share IPD: No